CLINICAL TRIAL: NCT02696798
Title: A Multicenter, Randomized, Double-Blind, Placebo- Controlled 16-Week Study Followed by Long-Term Evaluation of Efficacy and Safety of Ixekizumab (LY2439821) in TNFi-Experienced Patients With Radiographic Axial Spondyloarthritis
Brief Title: A Study of Ixekizumab (LY2439821) in TNF Inhibitor Experienced Participants With Radiographic Axial Spondyloarthritis
Acronym: COAST-W
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16179; I1F-MC-RHBW (Other: Eli Lilly and Company); 2015-003937-84 (EudraCT Number)
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Spondyloarthritis
Keywords: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylarthritis; Spondylitis, Ankylosing | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Q2W Ixekizumab (Experimental): Double Blind Period: Starting dose of 80 or 160 milligrams (mg) ixekizumab given subcutaneously (SC) at baseline followed by 80 mg ixekizumab given SC every two weeks (Q2W) to week 14.
  Extended Treatment Period: 80 mg ixekizumab given SC Q2W from week 16 to week 52.
  Interventions: Drug: Ixekizumab
- Q4W Ixekizumab (Experimental): Double Blind Period: Starting dose of 80 or 160 mg ixekizumab given SC at baseline followed by 80 mg ixekizumab given SC every four weeks (Q4W) to week 14.
  Extended Treatment Period: 80 mg ixekizumab given SC Q4W from week 16 to week 52.
  Interventions: Drug: Ixekizumab
- Placebo (Placebo Comparator): Double Blind Period: Placebo given SC Q2W to week 14.
  Extended Treatment Period: Starting dose of 160 mg ixekizumab given SC at week 16 followed by 80 mg ixekizumab given SC Q2W or Q4W from week 16 to week 52.
  Interventions: Drug: Ixekizumab; Drug: Placebo

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of ixekizumab in tumor necrosis factor (TNF) inhibitor-experienced participants with radiographic axial spondyloarthritis (rad-axSpA).

ELIGIBILITY:
Inclusion Criteria:

* Are ambulatory.
* Have an established diagnosis of radiographic axial spondyloarthritis (rad-xSpA) with sacroiliitis defined radiographically according to the modified New York criteria.
* Participants have a history of back pain ≥3 months with age at onset <45 years.
* Have had prior treatment with at least 1 and not more than 2 TNF inhibitors.
* Must have had an inadequate response to 2 or more NSAIDs at the therapeutic dose range for a total duration of at least 4 weeks OR have a history of intolerance to NSAIDs.
* Have a history of prior therapy for axSpa for at least 12 weeks prior to screening.

Exclusion Criteria:

* Have total ankylosis of the spine.
* Have never taken a TNF inhibitor medication or have taken more than 2.
* Have recently received a live vaccine within 12 weeks or have had a vaccination with Bacillus Calmette-Guerin (BCG) within the past year.
* Have an ongoing or serious infection within the last 12 weeks or evidence of active tuberculosis.
* Have a compromised immune system.
* Have any other serious and/or uncontrolled diseases.
* Have either a current diagnosis or a recent history of malignant disease.
* Have had major surgery within 8 weeks of baseline, or will require surgery during the study.
* Are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2019-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (88):
- United States (27):
  - Arizona Arthritis Research, PLC, Phoenix, Arizona
  - Rheumatology Center of San Diego, Escondido, California
  - Care Access Research - Huntington Beach, Huntington Beach, California
  - Desert Medical Advances, Palm Desert, California
  - Arthritis Assoc. & Osteoporosis Ctr of Colorado Springs, LLC, Colorado Springs, Colorado
  - Denver Arthritis Center, Denver, Colorado
  - Clinical Research Center of CT/NY, Danbury, Connecticut
  - Arthritis Rheumatic Disease Specialties, Aventura, Florida
  - Sarasota Arthritis Center, Sarasota, Florida
  - Marietta Rheumatology, Marietta, Georgia
  - St Luke's Clinic - Intermountain Orthopaedics, Boise, Idaho
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Center for Arthritis & Osteoporosis, Elizabethtown, Kentucky
  - Klein and Associates MD, PA, Cumberland, Maryland
  - Osteoporosis And Clinical Trial Center, Hagerstown, Maryland
  - Arthritis Consultants, St Louis, Missouri
  - The Center for Rheumatology, Albany, New York
  - Shanahan Rheumatology & Immunotherapy, Raleigh, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Articularis Healthcare Group, INC dba Columbia Arthritis Ctr, Columbia, South Carolina
  - Low Country Research Center, North Charleston, South Carolina
  - Univ of Texas Health Science Center - Houston, Houston, Texas
  - Southwest Rheumatology, P.A., Mesquite, Texas
  - Center for Arthritis and Rheumatic Diseases, PC, Chesapeake, Virginia
  - Arthritis Northwest Rheumatology, Spokane, Washington
  - Rheumatology and Immunotherapy Center, Franklin, Wisconsin
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Brazil (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiás
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Juiz de Fora
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., St. John's
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Trois-Rivières
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria
- Finland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyvinkää
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oulu
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Le Kremlin-Bicêtre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tours
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin, Germany
- Israel (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ashkelon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reggio Emilia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siena
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamagata
- Mexico (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexicali
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mérida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sneek
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Świdnik
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Puerto Rico (4):
  - Office: Perez-De Jesus, Amarilis, Caguas, PR
  - GCM Medical Group PSC, San Juan, PR
  - Mindful Medical Research, San Juan, PR
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elche
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- United Kingdom (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Basingstoke
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norwich
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Solihull
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stoke-on-Trent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wolverhampton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wythenshawe

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Reveille JD, Rudwaleit M, Rahman P, Maldonado-Cocco JA, Magrey M, Bolce R, Ng KJ, Gibble TH, Lisse J, Park SY, Kronbergs A, Navarro-Compan V. Does HLA-B27 Status Influence Ixekizumab Efficacy in Axial Spondyloarthritis? Results From the COAST-V, COAST-W, and COAST-X Trials. Rheumatol Ther. 2026 Feb;13(1):279-291. doi: 10.1007/s40744-025-00810-5. Epub 2025 Dec 19. PMID 41417207
- [Derived] Navarro-Compan V, Reveille JD, Rahman P, Maldonado-Cocco JA, Magrey M, Bolce R, Panni T, Kronbergs A, Rudwaleit M. Ixekizumab Improves Signs, Symptoms, and Quality of Life in Patients with Axial Spondyloarthritis Irrespective of Symptom Duration. Adv Ther. 2025 Sep;42(9):4706-4716. doi: 10.1007/s12325-025-03305-5. Epub 2025 Jul 22. PMID 40694276
- [Derived] Deodhar A, Poddubnyy D, Rahman P, Ermann J, Tomita T, Bolce R, Leage SL, Kronbergs A, Johnson C, Araujo J, Leung A, van der Heijde D. Long-Term Safety and Efficacy of Ixekizumab in Patients With Axial Spondyloarthritis: 3-year Data From the COAST Program. J Rheumatol. 2023 Aug;50(8):1020-1028. doi: 10.3899/jrheum.221022. Epub 2023 Feb 15. PMID 36792107
- [Derived] Ortolan A, Ramiro S, Ramonda R, van der Heijde D. External validation of the alternative Ankylosing Spondylitis Disease Activity Score in three randomized clinical trials of ixekizumab. Rheumatology (Oxford). 2023 Jun 1;62(6):2257-2261. doi: 10.1093/rheumatology/keac618. PMID 36282526
- [Derived] van der Horst-Bruinsma IE, de Vlam K, Walsh JA, Bolce R, Hunter T, Sandoval D, Zhu D, Geneus V, Soriano ER, Magrey M. Baseline Characteristics and Treatment Response to Ixekizumab Categorised by Sex in Radiographic and Non-radiographic Axial Spondylarthritis Through 52 Weeks: Data from Three Phase III Randomised Controlled Trials. Adv Ther. 2022 Jun;39(6):2806-2819. doi: 10.1007/s12325-022-02132-2. Epub 2022 Apr 16. PMID 35429281
- [Derived] Maksymowych WP, Bolce R, Gallo G, Seem E, Geneus VJ, Sandoval DM, Ostergaard M, Tada K, Baraliakos X, Deodhar A, Gensler LS. Ixekizumab in radiographic axial spondyloarthritis with and without elevated C-reactive protein or positive magnetic resonance imaging. Rheumatology (Oxford). 2022 Nov 2;61(11):4324-4334. doi: 10.1093/rheumatology/keac104. PMID 35188180
- [Derived] van der Heijde D, Ostergaard M, Reveille JD, Baraliakos X, Kronbergs A, Sandoval DM, Li X, Carlier H, Adams DH, Maksymowych WP. Spinal Radiographic Progression and Predictors of Progression in Patients With Radiographic Axial Spondyloarthritis Receiving Ixekizumab Over 2 Years. J Rheumatol. 2022 Mar;49(3):265-273. doi: 10.3899/jrheum.210471. Epub 2021 Dec 1. PMID 34853086
- [Derived] Deodhar AA, Mease PJ, Rahman P, Navarro-Compan V, Strand V, Hunter T, Bolce R, Leon L, Lauzon S, Marzo-Ortega H. Ixekizumab improves spinal pain, function, fatigue, stiffness, and sleep in radiographic axial Spondyloarthritis: COAST-V/W 52-week results. BMC Rheumatol. 2021 Sep 20;5(1):35. doi: 10.1186/s41927-021-00205-3. PMID 34538257
- [Derived] Dougados M, Wei JC, Landewe R, Sieper J, Baraliakos X, Van den Bosch F, Maksymowych WP, Ermann J, Walsh JA, Tomita T, Deodhar A, van der Heijde D, Li X, Zhao F, Bertram CC, Gallo G, Carlier H, Gensler LS; COAST-V and COAST-W Study Groups. Efficacy and safety of ixekizumab through 52 weeks in two phase 3, randomised, controlled clinical trials in patients with active radiographic axial spondyloarthritis (COAST-V and COAST-W). Ann Rheum Dis. 2020 Feb;79(2):176-185. doi: 10.1136/annrheumdis-2019-216118. Epub 2019 Nov 4. PMID 31685553
- [Derived] Mease P, Walsh JA, Baraliakos X, Inman R, de Vlam K, Wei JC, Hunter T, Gallo G, Sandoval D, Zhao F, Dong Y, Bolce R, Marzo-Ortega H. Translating Improvements with Ixekizumab in Clinical Trial Outcomes into Clinical Practice: ASAS40, Pain, Fatigue, and Sleep in Ankylosing Spondylitis. Rheumatol Ther. 2019 Sep;6(3):435-450. doi: 10.1007/s40744-019-0165-3. Epub 2019 Jun 28. PMID 31254223
- [Derived] Deodhar A, Poddubnyy D, Pacheco-Tena C, Salvarani C, Lespessailles E, Rahman P, Jarvinen P, Sanchez-Burson J, Gaffney K, Lee EB, Krishnan E, Santisteban S, Li X, Zhao F, Carlier H, Reveille JD; COAST-W Study Group. Efficacy and Safety of Ixekizumab in the Treatment of Radiographic Axial Spondyloarthritis: Sixteen-Week Results From a Phase III Randomized, Double-Blind, Placebo-Controlled Trial in Patients With Prior Inadequate Response to or Intolerance of Tumor Necrosis Factor Inhibitors. Arthritis Rheumatol. 2019 Apr;71(4):599-611. doi: 10.1002/art.40753. Epub 2019 Mar 8. PMID 30343531
- See also: Click here for more information about this study: A Study of Ixekizumab (LY2439821) in TNF Inhibitor Experienced Participants With Radiographic Axial Spondyloarthritis (COAST-W) — http://www.lillytrialguide.com/EN-us/studies/arthritis/rhbw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Blinded Treatment Dosing Period (Week 0 to Week 16), Extended Treatment Period (Week 16 to Week 52) followed by post-treatment follow-up period occurring from last treatment visit (week 52), or Early Termination Visit (ETV) up to a minimum of 12 weeks following that visit.
Pre-assignment Details: Participants who completed study were eligible to enroll into a long-term study (I1F-MC-RHBY [NCT03129100]) for up to 2 additional years. Participants who terminate study RHBW early or who do not enroll into Study RHBY will complete the Post-Treatment Follow-Up (PTFU) Period in study RHBW.
Groups:
- PBO/IXE: Blinded Treatment Dosing Period: Participants received placebo (PBO) every two weeks (Q2W) by subcutaneous (SC) injection during Week 0 to 16.
  Extended Treatment Period: Participants who received Placebo in blinded treatment period were re-randomized to receive ixekizumab (IXE) 80 mg every four weeks (Q4W) or 80 mg Q2W at a 1:1 ratio with starting dose of 160 mg.
  Post-treatment Follow-up Period: Participants did not receive any intervention during Follow-up period
- IXE80Q4W/IXE80Q4W: Blinded Treatment Dosing Period: Participants received starting dose of 80 or 160 mg ixekizumab given SC at baseline followed by 80 mg ixekizumab given SC every four weeks (Q4W) up to week 16.
  Extended Treatment Period: Participants received 80 mg ixekizumab given SC Q4W from week 16 to week 52.
  Post-treatment Follow-up Period: Participants did not receive any intervention during Follow-up period
- IXE80Q2W/IXE80Q2W: Blinded Treatment Dosing Period: Participants received starting dose of 80 or 160 milligrams (mg) ixekizumab given subcutaneously (SC) at baseline followed by 80 mg ixekizumab given SC every two weeks (Q2W) up to week 16.
  Extended Treatment Period: Participants received 80 mg ixekizumab given SC Q2W from week 16 to week 52.
  Post-treatment Follow-up Period: Participants did not receive any intervention during Follow-up period
Period: Blinded Treatment Dosing Period
Arm/Group | PBO/IXE | IXE80Q4W/IXE80Q4W | IXE80Q2W/IXE80Q2W
Started | 104 | 114 | 98
Completed | 93 | 99 | 90
Not Completed | 11 | 15 | 8
Not completed — Adverse Event | 2 | 9 | 2
Not completed — Death | 0 | 0 | 1
Not completed — Lack of Efficacy | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 3 | 4
Period: Extended Treatment Period
Arm/Group | PBO/IXE | IXE80Q4W/IXE80Q4W | IXE80Q2W/IXE80Q2W
Started | 93 | 98 (1 participant completed blinded treatment period and entered post-treatment followup period directly) | 90
Completed | 81 | 89 | 80
Not Completed | 12 | 9 | 10
Not completed — Adverse Event | 1 | 4 | 5
Not completed — Lack of Efficacy | 7 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 3
Period: Post-treatment Follow-up Period
Arm/Group | PBO/IXE | IXE80Q4W/IXE80Q4W | IXE80Q2W/IXE80Q2W
Started | 5 (Participants who terminate RHBW early or who didn't enroll into RHBY entered Follow-Up Period.) | 34 (Participants who terminate RHBW early or who didn't enroll into RHBY entered Follow-Up Period.) | 22 (Participants who terminate RHBW early or who didn't enroll into RHBY entered Follow-Up Period.)
Completed | 0 | 8 | 3
Not Completed | 5 | 26 | 19
Not completed — Adverse Event | 2 | 12 | 6
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Lack of Efficacy | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 8 | 12
Not completed — Physician Decision | 0 | 2 | 0
Not completed — No progressive improvement | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- PBO/IXE: Blinded Treatment Dosing Period: Participants received placebo every two weeks (Q2W) by subcutaneous (SC) injection during Week 0 to 16.
  Extended Treatment Period: Participants who received Placebo in blinded treatment period were re-randomized to receive ixekizumab 80 mg Q4W or 80 mg Q2W at a 1:1 ratio with starting dose of 160 mg.
  Post-treatment Follow-up Period: Participants did not receive any intervention during Follow-up period
  Participants did not receive any intervention during Follow-up period
- IXE80Q4W/IXE80Q4W: Blinded Treatment Dosing Period: Participants received starting dose of 80 or 160 mg ixekizumab given SC at baseline followed by 80 mg ixekizumab given SC every four weeks (Q4W) up to week 16.
  Extended Treatment Period: Participants received 80 mg ixekizumab given SC Q4W from week 16 to week 52.
  Post-treatment Follow-up Period: Participants did not receive any intervention during Follow-up period
  Participants did not receive any intervention during Follow-up period
- IXE80Q2W/IXE80Q2W: Blinded Treatment Dosing Period: Participants received starting dose of 80 or 160 milligrams (mg) ixekizumab given subcutaneously (SC) at baseline followed by 80 mg ixekizumab given SC every two weeks (Q2W) up to week 16.
  Extended Treatment Period: Participants received 80 mg ixekizumab given SC Q2W from week 16 to week 52.
  Post-treatment Follow-up Period: Participants did not receive any intervention during Follow-up period
  Participants did not receive any intervention during Follow-up period
- Total: Total of all reporting groups
Arm/Group | PBO/IXE | IXE80Q4W/IXE80Q4W | IXE80Q2W/IXE80Q2W | Total
Number analyzed (Participants) | 104 | 114 | 98 | 316
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (12.72) | 47.4 (13.36) | 44.2 (10.79) | 46.1 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 23 | 23 | 63
  Male | 87 | 91 | 75 | 253
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 32 | 35 | 100
  Not Hispanic or Latino | 63 | 70 | 53 | 186
  Unknown or Not Reported | 8 | 12 | 10 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 4 | 12
  Asian | 13 | 14 | 13 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 85 | 91 | 78 | 254
  More than one race | 1 | 2 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 1 | 2 | 4 | 7
  Argentina | 6 | 7 | 5 | 18
  United States | 14 | 14 | 12 | 40
  United Kingdom | 9 | 6 | 5 | 20
  Spain | 3 | 7 | 4 | 14
  Canada | 1 | 5 | 0 | 6
  South Korea | 12 | 11 | 11 | 34
  Netherlands | 1 | 2 | 0 | 3
  Finland | 0 | 3 | 2 | 5
  Brazil | 10 | 8 | 10 | 28
  Poland | 22 | 24 | 20 | 66
  Italy | 0 | 1 | 1 | 2
  Mexico | 13 | 13 | 13 | 39
  Israel | 5 | 5 | 6 | 16
  France | 7 | 5 | 5 | 17
  Germany | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an Assessment of Spondyloarthritis International Society 40 (ASAS40) Response
Description: ASAS40 is defined as improvement from baseline of greater than or equal to (>=) 40 % and absolute improvement from baseline of at least 2 units (range of 0 to 10) in at least 3 of the following 4 domains without any worsening in the remaining domain.
  1. Patient Global: How active was your spondylitis on average during the last week? score ranges 0 (not active) to 10 (very active).
  2. Spinal Pain: How much Pain of your spine due to Ankylosing spondylitis? score ranges 0 (no pain) to 10 (severe pain).
  3. Bath Ankylosing Spondylitis Functional Index (BASFI): Participant asked to rate the difficulty associated with 10 individual basic functional activities. Participant response was captured using Numeric Rating Scale (NRS) (range 0 to 10) with a higher score indicating worse function.
  4. Inflammation based on Q5 & Q6 mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) (mean of intensity & duration of stiffness): Score ranges from "0" (none) and "10" (very severe).
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo: Participants received placebo every 2 weeks (Q2W) by subcutaneous injection.
- 80 mg Q4W Ixekizumab: Participants received starting dose of 80 or 160 mg ixekizumab by SC injection at baseline followed by 80 mg ixekizumab given SC every four weeks (Q4W).
- 80 mg Q2W Ixekizumab: Participants received starting dose of 80 or 160 mg ixekizumab given SC injection at baseline followed by 80 mg ixekizumab given SC every two weeks (Q2W) to week 16.
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Percentage of participants | 12.5 | 25.4 | 30.6
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.017, Regression, Logistic; Odds Ratio (OR) = 2.41, 95% CI 2-sided [1.17 to 4.95]
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 3.06, 95% CI 2-sided [1.48 to 6.33]

2. Secondary Outcome: Percentage of Participants Achieving an ASAS20 Response
Description: ASAS20 response is defined as a ≥20% improvement and an absolute improvement from baseline of ≥1 units (range 0 to 10) in ≥3 of 4 domains, and no worsening of ≥20% and ≥1 unit (range 0 to 10) in the remaining domain.
  1. Patient Global: How active was your spondylitis on average during the last week? score ranges 0 (not active) to 10 (very active).
  2. Spinal Pain: How much Pain of your spine due to Ankylosing spondylitis? score ranges 0 (no pain) to 10 (severe pain).
  3. Bath Ankylosing Spondylitis Functional Index (BASFI): Participant asked to rate the difficulty associated with 10 individual basic functional activities. Participant response was captured using Numeric Rating Scale (NRS) (range 0 to 10) with a higher score indicating worse function.
  4. Inflammation based on Q5 & Q6 mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) (mean of intensity & duration of stiffness): Score ranges from "0" (none) and "10" (very severe).
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: Participants received placebo every 2 weeks by subcutaneous injection.
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Percentage of Participants | 29.8 | 48.2 | 46.9
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 2.20, 95% CI 2-sided [1.26 to 3.84]
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.013, Regression, Logistic; Odds Ratio (OR) = 2.08, 95% CI 2-sided [1.16 to 3.73]

3. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS)
Description: ASDAS is a composite index to assess disease activity in AS. The parameters used for the ASDAS (with CRP as acute phase reactant) are
  1. Total back pain
  2. Patient global
  3. Peripheral pain/swelling
  4. Duration of morning stiffness and
  5. CRP in mg/L. The ASDAScrp is calculated with the following equation: 0.121×total back pain+0.110×patient global+0.073×peripheral pain/swelling+0.058×duration of morning stiffness+0.579×Ln(CRP+1). (CRP is in mg/liter, the range of other variables is from 0(normal) to 10(very severe); Ln represents the natural logarithm). Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher scores indicated higher disease activity. Least Square (LS) mean was determined by mixed-model repeated measures (MMRM) with treatment, geographic region, baseline CRP status, number of prior tumor necrosis factor inhibitor (TNFi), baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Units on a scale | -0.11 (0.099) | -1.16 (0.094) | -1.13 (0.103)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.32 to -0.79], Standard Error of Mean 0.135
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-1.30 to -0.75], Standard Error of Mean 0.140

4. Secondary Outcome: Percentage of Participants Achieving Bath Ankylosing Spondylitis Disease Activity Index 50 (BASDAI50) Response
Description: The BASDAI is a participant-reported assessment consisting of 6 questions that relate to 5 major symptoms relevant to radiographic axial spondyloarthritis (rad-axSpA): 1) Fatigue, 2) Spinal pain, 3) Peripheral arthritis, 4) Enthesitis, 5) Intensity, and 6) Duration of morning stiffness. Participants need to score each item with a score from 0 to 10 (NRS). Total score is obtained from the average of symptom scores ranging 0 (no problem) to 10 (worst problem), with a higher score indicating more severe AS symptom. BASDAI50 represents an improvement of ≥50% of the BASDAI score from baseline.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Percentage of Participants | 9.6 | 21.9 | 23.5
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.015, Regression, Logistic; Odds Ratio (OR) = 2.65, 95% CI 2-sided [1.21 to 5.84]
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.010, Regression, Logistic; Odds Ratio (OR) = 2.90, 95% CI 2-sided [1.29 to 6.49]

5. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: The BASDAI is a participant-reported assessment consisting of 6 questions that relate to 5 major symptoms relevant to radiographic axial spondyloarthritis (rad-axSpA): 1) Fatigue, 2) Spinal pain, 3) Peripheral arthritis, 4) Enthesitis, 5) Intensity, and 6) Duration of morning stiffness. Participants need to score each item with a score from 0 to 10 (NRS). Total score is obtained from the average of symptom scores ranging 0 (no problem) to 10 (worst problem), with a higher score indicating more severe AS symptom. LSmean was determined by MMRM with factors for treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Units on a scale | -0.92 (0.212) | -2.17 (0.202) | -2.09 (0.221)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.24, 95% CI 2-sided [-1.81 to -0.67], Standard Error of Mean 0.291
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-1.76 to -0.57], Standard Error of Mean 0.301

6. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: The BASFI is a participant-reported assessment that establishes a participant's functional baseline and subsequent response to treatment. The BASFI is composed with 10 questions to assess the disease severity, including the first 8 questions regarding to functional anatomy related activities and the remaining 2 questions related to daily activities of AS participants. Participants respond to each question using an NRS scale (range 0 to 10). The BASFI score is the average of the 10 responses and has a possible minimum value of 0 and a possible maximum value of 10, with a higher score indicating worse function. LS mean was determined by MMRM with factors for treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Units on a scale | -0.64 (0.215) | -1.69 (0.205) | -1.92 (0.225)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.63 to -0.47], Standard Error of Mean 0.295
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-1.89 to -0.68], Standard Error of Mean 0.307

7. Secondary Outcome: Percentage of Participants Achieving ASDAS Inactive Disease
Description: ASDAS is a composite index to assess disease activity in AS. ASDAS Inactive Disease is defined as a score of <1.3.
  The parameters used for the ASDAS (with CRP as acute phase reactant) are
  1. Total back pain
  2. Patient global
  3. Peripheral pain/swelling
  4. Duration of morning stiffness and
  5. CRP in mg/L. The ASDAScrp is calculated with the following equation: 0.121×total back pain+0.110×patient global+0.073×peripheral pain/swelling+0.058×duration of morning stiffness+0.579×Ln(CRP+1). (CRP is in mg/liter, the range of other variables is from 0(normal) to 10(very severe); Ln represents the natural logarithm). Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher the score worse the disease activity.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Percentage of Participants | 1.0 | 3.5 | 5.1
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.242, Regression, Logistic; Odds Ratio (OR) = 3.73, 95% CI 2-sided [0.41 to 33.98]
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.127, Regression, Logistic; Odds Ratio (OR) = 5.42, 95% CI 2-sided [0.62 to 47.54]

8. Secondary Outcome: Percentage of Participants Achieving ASDAS <2.1
Description: ASDAS is a composite index to assess disease activity in AS. ASDAS <2.1 defines moderate disease activity.
  The parameters used for the ASDAS (with CRP as acute phase reactant) are
  1. Total back pain
  2. Patient global
  3. Peripheral pain/swelling
  4. Duration of morning stiffness and
  5. CRP in mg/L. The ASDAScrp is calculated with the following equation: 0.121×total back pain+0.110×patient global+0.073×peripheral pain/swelling+0.058×duration of morning stiffness+0.579×Ln(CRP+1). (CRP is in mg/liter, the range of other variables is from 0(normal) to 10(very severe); Ln represents the natural logarithm). Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher the score worse the disease activity.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Percentage of Participants | 4.8 | 17.5 | 16.3
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 4.22, 95% CI 2-sided [1.50 to 11.86]
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 4.52, 95% CI 2-sided [1.55 to 13.18]

9. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores
Description: The SF-36 is a 36-item participant administered measure designed to be a short, multipurpose assessment of health in the areas of physical functioning, role - physical, role - emotional, bodily pain, vitality, social functioning, mental health, and general health. The 2 overarching domains of mental well- being and physical well-being are captured by the Mental Component Summary and Physical Component Summary scores. T-scores are used for analysis. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. LSmean was determined by MMRM with factors for treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Units on a scale
  SF-36 MCS | 2.7410 (0.9452) | 3.5099 (0.9074) | 3.6514 (0.9921)
  SF-36 PCS | 1.3638 (0.8146) | 6.5785 (0.7763) | 6.1223 (0.8465)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; MCS; Test type: Superiority; p = 0.550, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.7689, 95% CI 2-sided [-1.7629 to 3.3007], Standard Error of Mean 1.2863
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; MCS; Test type: Superiority; p = 0.495, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.9104, 95% CI 2-sided [-1.7151 to 3.5360], Standard Error of Mean 1.3338
Statistical Analysis 3: Comparison: Placebo vs 80 mg Q4W Ixekizumab; PCS; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = 5.2147, 95% CI 2-sided [3.0204 to 7.4090], Standard Error of Mean 1.1149
Statistical Analysis 4: Comparison: Placebo vs 80 mg Q2W Ixekizumab; PCS; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = 4.7585, 95% CI 2-sided [2.4940 to 7.0230], Standard Error of Mean 1.1505

10. Secondary Outcome: Change From Baseline in ASAS Health Index (ASAS HI)
Description: The ASAS Health Index (ASAS HI) is a disease specific health-index instrument designed to assess the impact of interventions for SpA, including axSpA. The 17 item instrument has scores ranging from 0 (good Health) to 17 (poor Health). Each item consists of 1 question that the patient needs to respond to with either "I agree" (score 1) or "I do not agree (score 0)." A score of "1" is given where the item is affirmed, indicating adverse health. All item scores are summed to give a total score or index. LS mean was determined by MMRM with treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Units on a scale | -0.89 (0.338) | -1.92 (0.322) | -1.58 (0.352)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.026, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-1.94 to -0.13], Standard Error of Mean 0.460
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.149, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.63 to 0.25], Standard Error of Mean 0.477

11. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) of the Spine (Ankylosing Spondylitis Spinal Magnetic Resonance Imaging [ASSpiMRI] - Berlin Score)
Description: The study used MRI with fat-saturating techniques such as short tau inversion recovery (STIR) to look for the presence of bone marrow edema. The Berlin modification of Ankylosing Spondylitis spine MRI score for activity (ASspiMRI) scoring technique assesses inflammation in each of the 23 disco-vertebral units (DVU) of the spine (from C2 to S1), capturing bone marrow edema. Scores for each DVU range from 0-3 (0=normal; 1=minor bone marrow edema [less than or equal to 25% of DVU; 3=severe bone marrow edema (more that 50% of DVU)]. The composite score ranges from 0 to 69, with higher scores reflecting worse disease.LS mean was determined by analysis of covariance (ANCOVA) with treatment, geographic region, baseline CRP status, number of prior TNF inhibitors used and baseline value as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and week 16 ASSpiMRI score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 46 | 49 | 45
Units on a scale | 1.03 (0.379) | -0.92 (0.373) | -1.14 (0.414)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = -1.95, 95% CI 2-sided [-3.0 to -0.9], Standard Error of Mean 0.512
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = -2.17, 95% CI 2-sided [-3.2 to -1.1], Standard Error of Mean 0.534

12. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) of the Spine (Spondyloarthritis Research Consortium of Canada [SPARCC] Score)
Description: MRI score of spine was assessed using SPARCC method. All 23 disco-vertebral units (DVU) of the spine (from C2 to S1) were scored for bone marrow edema. A single DVU has 18 scoring units, and each has score of 0 or 1, bringing the maximum total score to 414, the sum ranges from 0 to 414 with higher scores reflecting worse disease. Scoring was performed by central readers. LS mean was determined by ANCOVA with factors for treatment, geographic region, baseline CRP status, number of prior TNF inhibitors used and baseline value.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and week 16 SPARCC MRI score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 46 | 49 | 45
Units on a scale | 3.29 (1.402) | -2.99 (1.384) | -3.97 (1.534)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.001, ANCOVA; LS Mean Difference (Final Values) = -6.29, 95% CI 2-sided [-10.0 to -2.5], Standard Error of Mean 1.896
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = -7.27, 95% CI 2-sided [-11.2 to -3.4], Standard Error of Mean 1.978

13. Secondary Outcome: Change From Baseline in the Measure of High Sensitivity C-Reactive Protein (CRP)
Description: High sensitivity CRP is the measure of acute phase reactant. It was measured with a high sensitivity assay at the central laboratory to help assess the effect of ixekizumab on disease activity. High sensitivity CRP is a sensitive laboratory assay for serum levels of C-Reactive Protein, which is a biomarker of inflammation. LS mean was determined by MMRM with treatment, geographic region, baseline CRP status, number of prior TNFi, visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: milligram per liter (mg/L)
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
milligram per liter (mg/L) | 9.719 (2.7383) | -11.096 (2.6190) | -8.121 (2.8829)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -20.816, 95% CI 2-sided [-28.187 to -13.444], Standard Error of Mean 3.7463
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -17.841, 95% CI 2-sided [-25.518 to -10.163], Standard Error of Mean 3.9018

14. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI)
Description: BASMI is a combined index comprising of 5 clinical measurements of spinal mobility in patients with radiographic axial spondyloarthritis (rad-axSpA).
  1. Lateral Spinal Flexion
  2. Tragus-to-wall distance
  3. Lumbar Flexion (modified Schober)
  4. Maximal intermalleolar distance and
  5. Cervical rotation. The BASMI linear result is the average of the 5 assessments and ranges from 0 to 10. The higher the BASMI score the more severe the patient's limitation of movement due to their AS. LS mean was determined by MMRM with treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Units on a scale | -0.046 (0.0939) | -0.349 (0.0897) | -0.217 (0.0981)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.018, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.304, 95% CI 2-sided [-0.555 to -0.053], Standard Error of Mean 0.1275
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.194, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.172, 95% CI 2-sided [-0.431 to 0.088], Standard Error of Mean 0.1319

15. Secondary Outcome: Change From Baseline in Chest Expansion
Description: Chest expansion is the difference, in centimeter (cm), between the circumference of the chest in maximal inspiration and maximal expiration. While patients have their hands resting on or behind the head, the assessor will measure the chest encircled length by centimeter (cm) at the fourth intercostal level anteriorly. Two tries were recorded. The better measurement (larger difference) of 2 tries (in centimeters) was used for analyses. LS mean was determined by MMRM with treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: centimeter(cm)
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
centimeter(cm) | 0.04 (0.644) | 1.27 (0.618) | 0.27 (0.655)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.170, Mixed Models Analysis; LS Mean Difference (Final Values) = 1.23, 95% CI 2-sided [-0.53 to 2.99], Standard Error of Mean 0.893
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.800, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-1.57 to 2.04], Standard Error of Mean 0.916

16. Secondary Outcome: Change From Baseline in Occiput to Wall Distance
Description: The participant is to make a maximum effort to touch the head against the wall when standing with heels and back against the wall (occiput). Then the distance from occiput to wall is measured. Two tries will be recorded. The better (smaller) measurement of 2 tries (in centimeters) will be used for analyses. LS mean was determined by MMRM with factors for treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
cm | 0.35 (0.384) | 0.03 (0.365) | -0.65 (0.399)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.547, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-1.34 to 0.71], Standard Error of Mean 0.521
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.064, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-2.06 to 0.06], Standard Error of Mean 0.538

17. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES)
Description: The MASES is an index used to measure the severity of enthesitis. The MASES assesses 13 sites for enthesitis using a score of "0" for no activity or "1" for activity. Sites assessed include costochondral 1 (right/left), costochondral 7 (right/left), spinal iliaca anterior superior (right/left), crista iliaca (right/left), spina iliaca posterior (right/left), processus spinosus L5, and Achilles tendon proximal insertion (right/left). The MASES is the sum of all site scores (range 0 to 13); higher scores indicate more severe enthesitis. LS mean was determined by MMRM with treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline MASES score > 0.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 69 | 82 | 74
Units on a scale | -1.9 (0.43) | -1.8 (0.40) | -2.2 (0.42)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.861, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.0 to 1.3], Standard Error of Mean 0.58
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.626, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.4 to 0.9], Standard Error of Mean 0.59

18. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Score
Description: The SPARCC enthesitis is an index used to measure the severity of enthesitis. The SPARCC assesses 16 sites for enthesitis using a score of "0" for no activity or "1" for activity. Sites assessed include Medial epicondyle (left/right [L/R]), Lateral epicondyle (L/R), Supraspinatus insertion into greater tuberosity of humerus (L/R), Greater trochanter (L/R), Quadriceps insertion into superior border of patella (L/R), Patellar ligament insertion into inferior pole of patella or tibial tubercle (L/R), Achilles tendon insertion into calcaneum (L/R), and Plantar fascia insertion into calcaneum (L/R). The SPARCC is the sum of all site scores (range 0 to 16). Higher scores indicate more severe enthesitis. LS mean was determined by MMRM with treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline SPARCC Enthesitis score > 0.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 60 | 78 | 64
Units on a scale | -1.9 (0.44) | -2.3 (0.40) | -1.8 (0.45)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.504, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.6 to 0.8], Standard Error of Mean 0.59
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.860, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.1 to 1.3], Standard Error of Mean 0.62

19. Secondary Outcome: Change From Baseline in Severity of Peripheral Arthritis by Tender Joint Count (TJC) Scores
Description: The number of tender and painful joints was determined by examination of 46 joints (23 joints on each side of the body). The 46 joints were assessed and classified as tender or not tender. Sum of all joints checked to be tender/painful divided by number of evaluable joints which was multiplied by 46 to obtain TJC score. The scores ranges from 0 (no tender/painful joints) to 46 (all joints tender/painful). LS mean was determined by MMRM with treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline TJC > 0.
Measure: Least Squares Mean (Standard Error); unit: Tender Joint Count
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 65 | 85 | 69
Tender Joint Count | -3.9 (0.79) | -4.8 (0.69) | -5.0 (0.79)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.362, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-3.0 to 1.1], Standard Error of Mean 1.03
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.303, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.3 to 1.0], Standard Error of Mean 1.08

20. Secondary Outcome: Change From Baseline in Severity of Peripheral Arthritis by Swollen Joint Count (SJC) Scores
Description: The number of swollen joints was determined by examination of 44 joints (22 joints on each side of the body). The 44 joints were assessed and classified as swollen or not swollen. Sum of all joints checked to be swollen divided by number of evaluable joints which was multiplied by 44 to obtain SJC score. The SJC score ranges from 0 (no swollen joints) to 44 (all joints swollen). LS mean was determined by MMRM with treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline SJC > 0.
Measure: Least Squares Mean (Standard Error); unit: Swollen Joint Count
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 45 | 48 | 44
Swollen Joint Count | -2.4 (0.51) | -2.6 (0.49) | -3.0 (0.54)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.813, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.5 to 1.2], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.410, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.0 to 0.8], Standard Error of Mean 0.71

21. Secondary Outcome: Percentage of Participants With Anterior Uveitis
Description: Anterior uveitis is an inflammation of the middle layer of the eye. which includes the iris (colored part of the eye) and the adjacent tissue, known as the ciliary body.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Percentage of Participants | 0 | 1.8 | 3.1

22. Secondary Outcome: Change From Baseline in the Fatigue Numeric Rating Scale (NRS) Score
Description: The fatigue severity NRS is a participant administered single-item 11-point horizontal scale anchored at 0 and 10, with 0 representing "no fatigue" and 10 representing "as bad as you can imagine". Participants rate their fatigue (feeling tired or worn out) by circling the 1 number that describes their worst level of fatigue during the previous 24 hours. LS mean was determined by MMRM with treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Units on a scale | -0.7 (0.24) | -2.0 (0.23) | -1.7 (0.25)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-1.9 to -0.6], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.005, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.6 to -0.3], Standard Error of Mean 0.34

23. Secondary Outcome: Change From Baseline in the Jenkins Sleep Evaluation Questionnaire (JSEQ)
Description: The Jenkins Sleep Evaluation Questionnaire (JSEQ) is a 4 item scale designed to estimate sleep problems in clinical research. The JSEQ assesses the frequency of sleep disturbance in 4 categories: 1) trouble falling asleep, 2) waking up several times during the night, 3) having trouble staying asleep (including waking up far too early), and 4) waking up after the usual amount of sleep feeling tired and worn out. Patients report the numbers of days they experience each of these problems in the past month on a 6 point Likert Scale ranging from 0 = "no days" to 5 = "22-30 days. The total JSEQ score ranges from 0 to 20, with higher scores indicating greater sleep disturbance. LS mean was determined by MMRM with treatment, geographic region, baseline CRP status, number of prior TNFi, baseline value, visit, baseline value-by-visit and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 114 | 98
Units on a scale | -1.8 (0.50) | -3.0 (0.48) | -2.4 (0.52)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Test type: Superiority; p = 0.088, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.5 to 0.2], Standard Error of Mean 0.68
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Test type: Superiority; p = 0.366, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.0 to 0.7], Standard Error of Mean 0.70

24. Secondary Outcome: Change From Baseline in the Work Productivity Activity Impairment Spondyloarthritis (WPAI-SpA) Scores
Description: The WPAI-SpA consists of 6 questions to determine employment status, hours missed from work because of SpA, hours missed from work for other reasons, hours actually worked, the degree to which SpA affected work productivity while at work, and the degree to which SpA affected activities outside of work. The WPAI-SpA has been validated in the rad-axSpA patient population. Four scores are derived: percentage of absenteeism, percentage of presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism, and percentage of impairment in activities performed outside of work. The computed percentage range for each sub-scale was from 0-100, with higher scores indicating greater impairment and less productivity. LS mean was determined by ANCOVA with treatment, geographic region, baseline CRP status, number of prior TNFi and baseline value as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and week 16 WPAI-SpA score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 99 | 112 | 96
Units on a scale
  Overall Work Impairment Score: number analyzed (Participants) | 54 | 44 | 43
  Overall Work Impairment Score | -9.84 (3.733) | -20.97 (4.016) | -23.50 (4.225)
  Percentage of Activity Impairment | -10.1 (2.60) | -16.5 (2.44) | -18.4 (2.74)
Statistical Analysis 1: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Overall Work Impairment Score; Test type: Superiority; p = 0.038, ANCOVA; LS Mean Difference (Final Values) = -11.13, 95% CI 2-sided [-21.65 to -0.60], Standard Error of Mean 5.323
Statistical Analysis 2: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Overall Work Impairment Score; Test type: Superiority; p = 0.012, ANCOVA; LS Mean Difference (Final Values) = -13.66, 95% CI 2-sided [-24.23 to -3.10], Standard Error of Mean 5.341
Statistical Analysis 3: Comparison: Placebo vs 80 mg Q4W Ixekizumab; Percentage of Activity Impairment; Test type: Superiority; p = 0.071, ANCOVA; LS Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-13.2 to 0.5], Standard Error of Mean 3.50
Statistical Analysis 4: Comparison: Placebo vs 80 mg Q2W Ixekizumab; Percentage of Activity Impairment; Test type: Superiority; p = 0.024, ANCOVA; LS Mean Difference (Final Values) = -8.3, 95% CI 2-sided [-15.5 to -1.1], Standard Error of Mean 3.65

25. Secondary Outcome: Change From Baseline in ASAS-Nonsteroidal Anti-Inflammatory Drug (NSAID) Score
Description: ASAS-NSAID score is used to present the NSAID intake by considering the type of NSAID, the total dose, & the number of days taking NSAID during a period of interest (PI). For NSAID equivalent scoring system, range is from 0 to 100, higher the score greated the NSAID intake. ASAS-NSAID score= (equivalent NSAID score) x (days of intake during PI) x (days per week)/(PI in days).
Time Frame: Baseline, Week 52
Population: Participants from extended treatment period who had NSAID Intake at baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- PBO/IXE: Blinded Treatment Dosing Period: Participants received placebo every two weeks (Q2W) by subcutaneous (SC) injection during Week 0 to 16.
  Extended Treatment Period: Participants who received Placebo in blinded treatment period were re-randomized to receive ixekizumab 80 mg Q4W or 80 mg Q2W at a 1:1 ratio.
- IXE80Q4W/IXE80Q4W: Blinded Treatment Dosing Period: Participants received starting dose of 80 or 160 mg ixekizumab given SC at baseline followed by 80 mg ixekizumab given SC every four weeks (Q4W) up to week 16.
  Extended Treatment Period: Participants received 80 mg ixekizumab given SC Q4W from week 16 to week 52.
- IXE80Q2W/IXE80Q2W: Blinded Treatment Dosing Period: Participants received starting dose of 80 or 160 milligrams (mg) ixekizumab given subcutaneously (SC) at baseline followed by 80 mg ixekizumab given SC every two weeks (Q2W) up to week 16.
  Extended Treatment Period: Participants received 80 mg ixekizumab given SC Q2W from week 16 to week 52.
Arm/Group | PBO/IXE | IXE80Q4W/IXE80Q4W | IXE80Q2W/IXE80Q2W
Number analyzed (Participants) | 69 | 71 | 58
Units on a scale | -9.84 (34.435) | -5.52 (19.553) | -2.33 (24.019)

26. Secondary Outcome: Percentage of Participants With Anti-Ixekizumab Antibodies
Description: A treatment emergent - antidrug antibody (TE-ADA) positive patient is defined as: a) a patient with a >= 4-fold increase over a positive baseline antibody titer; or b) for a negative baseline titer, a patient with an increase from the baseline to a level of >= 1:10. Percentage was calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-ixekizumab antibodies / number of evaluable participants * 100%.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 80 mg Q4W Ixekizumab | 80 mg Q2W Ixekizumab
Number analyzed (Participants) | 104 | 113 | 98
Percentage of Participants | 2.9 | 7.1 | 4.1

27. Secondary Outcome: Pharmacokinetics (PK): Trough Ixekizumab Concentration at Steady State (Ctrough ss)
Description: Pharmacokinetics (PK): Steady-state trough serum concentration of Ixekizumab at week 16.
Time Frame: Week 16
Population: All randomized participants who received study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliters (µg/mL)
Groups:
- 80 mg Q4W Ixekizumab (Starting Dose 80 mg): Participants received 80 mg of Ixekizumab every four weeks by subcutaneous injection.
- 80 mg Q4W Ixekizumab (Starting Dose 160 mg): Participants received 160 mg ixekizumab at baseline followed by 80 mg ixekizumab given SC every four weeks by subcutaneous injection.
- 80 mg Q2W Ixekizumab (Starting Dose 80 mg): Participants received 80 mg ixekizumab every two weeks by subcutaneous injection.
- 80 mg Q2W Ixekizumab (Starting Dose 160 mg): Participants received starting dose of 160 mg ixekizumab at baseline followed by 80 mg ixekizumab every two weeks by subcutaneous injection.
Arm/Group | 80 mg Q4W Ixekizumab (Starting Dose 80 mg) | 80 mg Q4W Ixekizumab (Starting Dose 160 mg) | 80 mg Q2W Ixekizumab (Starting Dose 80 mg) | 80 mg Q2W Ixekizumab (Starting Dose 160 mg)
Number analyzed (Participants) | 60 | 54 | 48 | 50
Microgram per milliliters (µg/mL) | 2.10 (106) | 2.47 (101) | 6.27 (158) | 8.52 (50)

ADVERSE EVENTS:
Time Frame: Up To 76 Weeks
Description: All randomized participants. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Groups:
- 80 mg Q2W Ixekizumab-Blinded Treatment Period: Participants received starting dose of 80 or 160 milligrams (mg) ixekizumab given subcutaneously (SC) at baseline followed by 80 mg ixekizumab given SC every two weeks (Q2W) up to week 16.
- 80 mg Q4W Ixekizumab-Blinded Treatment Period: Participants received starting dose of 80 or 160 mg ixekizumab given SC at baseline followed by 80 mg ixekizumab given SC every four weeks (Q4W) up to week 16.
- PBO-Blinded Treatment Period: Participants received placebo every two weeks (Q2W) by subcutaneous (SC) injection during Week 0 to 16.
- IXE80Q2W/IXE80Q2W-Extended Treatment Period: Participants received 80 mg ixekizumab given SC Q2W from week 16 to week 52.
- IXE80Q4W/IXE80Q4W-Extended Treatment Period; PBO/IXE-Extended Treatment Period: Participants received 80 mg ixekizumab given SC Q4W from week 16 to week 52.
- IXE80Q2W-Follow-up Period; IXE80Q4W-Follow-up Period; PBO-Follow-up Period: Participants did not receive any intervention during post-treatment follow-up period.
Arm/Group | 80 mg Q2W Ixekizumab-Blinded Treatment Period | 80 mg Q4W Ixekizumab-Blinded Treatment Period | PBO-Blinded Treatment Period | IXE80Q2W/IXE80Q2W-Extended Treatment Period | IXE80Q4W/IXE80Q4W-Extended Treatment Period | PBO/IXE-Extended Treatment Period | IXE80Q2W-Follow-up Period | IXE80Q4W-Follow-up Period | PBO-Follow-up Period
All-Cause Mortality (participants affected / at risk) | 1/98 | 0/114 | 0/104 | 0/90 | 0/98 | 0/93 | 0/22 | 0/34 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/98 | 4/114 | 5/104 | 1/90 | 2/98 | 6/93 | 1/22 | 2/34 | 0/5
Other Adverse Events (participants affected / at risk) | 25/98 | 25/114 | 12/104 | 26/90 | 19/98 | 19/93 | 1/22 | 3/34 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 80 mg Q2W Ixekizumab-Blinded Treatment Period (N=98) | 80 mg Q4W Ixekizumab-Blinded Treatment Period (N=114) | PBO-Blinded Treatment Period (N=104) | IXE80Q2W/IXE80Q2W-Extended Treatment Period (N=90) | IXE80Q4W/IXE80Q4W-Extended Treatment Period (N=98) | PBO/IXE-Extended Treatment Period (N=93) | IXE80Q2W-Follow-up Period (N=22) | IXE80Q4W-Follow-up Period (N=34) | PBO-Follow-up Period (N=5)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drop attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meralgia paraesthetica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 80 mg Q2W Ixekizumab-Blinded Treatment Period (N=98) | 80 mg Q4W Ixekizumab-Blinded Treatment Period (N=114) | PBO-Blinded Treatment Period (N=104) | IXE80Q2W/IXE80Q2W-Extended Treatment Period (N=90) | IXE80Q4W/IXE80Q4W-Extended Treatment Period (N=98) | PBO/IXE-Extended Treatment Period (N=93) | IXE80Q2W-Follow-up Period (N=22) | IXE80Q4W-Follow-up Period (N=34) | PBO-Follow-up Period (N=5)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 6 (6) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 8 (21) | 3 (5) | 1 (1) | 5 (14) | 2 (2) | 3 (9) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 5 (5) | 2 (2) | 4 (4) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 9 (12) | 3 (3) | 8 (10) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/23 (0) | 0/23 (0) | 0/17 (0) | 0/22 (0) | 0/17 (0) | 1/16 (1) | 0/4 (0) | 0/9 (0) | 0/1 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (8) | 4 (4) | 2 (2) | 4 (4) | 4 (5) | 1 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 5 (5) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0/23 (0) | 0/23 (0) | 0/17 (0) | 0/22 (0) | 1/17 (1) | 0/16 (0) | 0/4 (0) | 0/9 (0) | 0/1 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0/23 (0) | 0/23 (0) | 0/17 (0) | 0/22 (0) | 1/17 (1) | 0/16 (0) | 0/4 (0) | 0/9 (0) | 0/1 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT02696798/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT02696798/SAP_001.pdf